CLINICAL TRIAL: NCT05738369
Title: The Effect of Probiotic Lozenges on White Spot Lesion Development in Orthodontic Patients: Prospective Randomized Controlled Trial
Brief Title: The Effect of Probiotic Lozenges on White Spot Lesion Development in Orthodontic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JUST20220097
Record Dates: First submitted 2023-02-04; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: White Spot Lesion
Keywords: White spot lesions, Probiotic lozenges, QLF

STUDY DESIGN:
Intervention Model Description: Three arm parallel design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigated supplements were provided to the participants by a research assistant. The participants in the negative control group, however, were not blinded because they did not receive any supplements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic (Experimental): Participants received treatment with Biogaia L. reuteri Prodentis® lozenges
  Interventions: Dietary Supplement: Biogaia L. reuteri Prodentis® lozenges
- Sugar free lozenges (Placebo Comparator): Participants received Hersheyland Ice Breakers Mints sugar free lozenges
  Interventions: Dietary Supplement: Hersheyland Ice Breakers Mints sugar free lozenges
- Negative control (No Intervention): Participants received no lozenges or supplements

INTERVENTIONS:
Dietary Supplement: Biogaia L. reuteri Prodentis® lozenges — Participants were instructed to use the lozenges twice daily after brushing their teeth; once in the morning and once in the evening
  Arms: Probiotic
Dietary Supplement: Hersheyland Ice Breakers Mints sugar free lozenges — Hersheyland Ice Breakers Mints sugar free lozenges
  Arms: Sugar free lozenges

SUMMARY:
The goal of this randomized clinical trial was to investigate the effect of probiotic lozenges on the development of white spot lesions (WSLs) compared to a positive control, and no treatment.

DETAILED DESCRIPTION:
Background: Recently, the use of probiotics has emerged as a treatment for prevention of oral cavity diseases including periodontal problems, and initial caries. The objectives of this prospective randomized clinical trial was to investigate the effect of probiotic lozenges on the development of white spot lesions (WSLs) compared to a positive control, and no treatment. Methods: Quantitative light induced fluorescence (QLF) images were taken for three randomly allocated groups (intervention group, n=23; positive control, n=23; negative control, n=24) of patients undergoing orthodontic treatment in three separate occasions (T0: before the start of study; T1: at 6 weeks later; T2: at 3 months after the commencement of the study). Subjects in the intervention group were instructed to take one probiotic lozenge containing two strains of Lactobacillus reuteri twice daily. Sugar-free lozenges were used in the positive control group and no lozenges for the negative control group. The QLF images were analyzed using a dedicated software in order to quantitatively analyze each tooth. The primary outcomes measured were the number of newly developed lesions in each group, lesion area and amount of mineral loss (ΔF). Means and standard deviations were calculated using the Statistical Package for the Social Science (SPSS version 28, Chicago, IL, USA). Split plot ANOVA (SPANOVA) test for repeated measures was used to check differences within and between the three groups regarding lesion area and ΔF. To check which group is different from the others, Tukey's test was used.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients from both sexes
* Having full fixed orthodontic appliances with expected remaining treatment duration of at least 6 months
* Optimum oral hygiene
* Maximum of 3 restored teeth
* Absence of defective enamel formation in the form of hypocalcification or hypoplasia

Exclusion Criteria:

* Patients with poor oral hygiene
* Defective enamel
* Extensive restorations
* Gingival hyperplasia
* Salivary glands diseases
* Smoking, alcohol consumption, mouth wash use, antibiotic or probiotic intake in the last 3 months.

Ages: 17 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of white spot lesions (WSL) | 3 months
  Number of newly developed white spot lesions
Lesion area | 3 months
  Surface area of the WSL (in pixels)
ΔF% | 3 months
  Average lesion fluorescence loss (ΔF%) reflecting mineral loss in percent.

SECONDARY OUTCOMES:
ΔFMax (%) | 3 months
  Deepest point in the lesion
ΔR30 (%) | 3 months
  Amount of plaque present

CONTACTS AND LOCATIONS:
Overall Officials: Susan Al-Khateeb, Principal Investigator — Faculty of Dentistry/Jordan University of Science and Technology
Locations (1):
- Postgraduate Dental Teaching Clinics/JUST, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
Data will be available upon request

REFERENCES:
- [Background] Gorelick L, Geiger AM, Gwinnett AJ. Incidence of white spot formation after bonding and banding. Am J Orthod. 1982 Feb;81(2):93-8. doi: 10.1016/0002-9416(82)90032-x. PMID 6758594
- [Background] Boersma JG, van der Veen MH, Lagerweij MD, Bokhout B, Prahl-Andersen B. Caries prevalence measured with QLF after treatment with fixed orthodontic appliances: influencing factors. Caries Res. 2005 Jan-Feb;39(1):41-7. doi: 10.1159/000081655. PMID 15591733
- [Background] 3. Øgaard, B. White spot lesions during orthodontic treatment: mechanisms and fluoride preventive aspects. Semin Orthod. 2008; 14: 183-193). WB Saunders.
- [Background] van Loveren C, Duggal MS. Experts' opinions on the role of diet in caries prevention. Caries Res. 2004;38 Suppl 1:16-23. doi: 10.1159/000074358. PMID 14685020
- [Background] Moynihan P, Petersen PE. Diet, nutrition and the prevention of dental diseases. Public Health Nutr. 2004 Feb;7(1A):201-26. doi: 10.1079/phn2003589. PMID 14972061
- [Background] Anusha RL, Umar D, Basheer B, Baroudi K. The magic of magic bugs in oral cavity: Probiotics. J Adv Pharm Technol Res. 2015 Apr-Jun;6(2):43-7. doi: 10.4103/2231-4040.154526. PMID 25878972
- [Background] 7. FAO/WHO. Evaluation of health and nutritional properties of powder milk and live lactic acid bacteria. Food and Agriculture Organization of the United Nations and World Health Organization Expert Consultation Report. 2001; 1-34.
- [Background] Flichy-Fernandez AJ, Alegre-Domingo T, Penarrocha-Oltra D, Penarrocha-Diago M. Probiotic treatment in the oral cavity: an update. Med Oral Patol Oral Cir Bucal. 2010 Sep 1;15(5):e677-80. doi: 10.4317/medoral.15.e677. PMID 20173706
- [Background] Doron S, Gorbach SL. Probiotics: their role in the treatment and prevention of disease. Expert Rev Anti Infect Ther. 2006 Apr;4(2):261-75. doi: 10.1586/14787210.4.2.261. PMID 16597207
- [Background] Jose JE, Padmanabhan S, Chitharanjan AB. Systemic consumption of probiotic curd and use of probiotic toothpaste to reduce Streptococcus mutans in plaque around orthodontic brackets. Am J Orthod Dentofacial Orthop. 2013 Jul;144(1):67-72. doi: 10.1016/j.ajodo.2013.02.023. PMID 23810047
- [Background] Galofre M, Palao D, Vicario M, Nart J, Violant D. Clinical and microbiological evaluation of the effect of Lactobacillus reuteri in the treatment of mucositis and peri-implantitis: A triple-blind randomized clinical trial. J Periodontal Res. 2018 Jun;53(3):378-390. doi: 10.1111/jre.12523. Epub 2018 Jan 19. PMID 29352461
- [Background] Guerrieri A, Gaucher C, Bonte E, Lasfargues JJ. Minimal intervention dentistry: part 4. Detection and diagnosis of initial caries lesions. Br Dent J. 2012 Dec;213(11):551-7. doi: 10.1038/sj.bdj.2012.1087. PMID 23222326
- [Background] Ando M, Hall AF, Eckert GJ, Schemehorn BR, Analoui M, Stookey GK. Relative ability of laser fluorescence techniques to quantitate early mineral loss in vitro. Caries Res. 1997;31(2):125-31. doi: 10.1159/000262387. PMID 9118184
- [Background] Al-Khateeb S, Forsberg CM, de Josselin de Jong E, Angmar-Mansson B. A longitudinal laser fluorescence study of white spot lesions in orthodontic patients. Am J Orthod Dentofacial Orthop. 1998 Jun;113(6):595-602. doi: 10.1016/s0889-5406(98)70218-5. PMID 9637561
- [Background] Pretty IA, Hall AF, Smith PW, Edgar WM, Higham SM. The intra- and inter-examiner reliability of quantitative light-induced fluorescence (QLF) analyses. Br Dent J. 2002 Jul 27;193(2):105-9. doi: 10.1038/sj.bdj.4801496. PMID 12199119
- [Background] Al-Khateeb S, Exterkate RA, de Josselin de Jong E, Angmar-Mansson B, ten Cate JM. Light-induced fluorescence studies on dehydration of incipient enamel lesions. Caries Res. 2002 Jan-Feb;36(1):25-30. doi: 10.1159/000057586. PMID 11961326
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] Albhaisi Z, Al-Khateeb SN, Abu Alhaija ES. Enamel demineralization during clear aligner orthodontic treatment compared with fixed appliance therapy, evaluated with quantitative light-induced fluorescence: A randomized clinical trial. Am J Orthod Dentofacial Orthop. 2020 May;157(5):594-601. doi: 10.1016/j.ajodo.2020.01.004. PMID 32354432
- [Background] 20. Dahlberg, G. Statistical methods for medical and biological students. Statistical Methods for Medical and Biological Students. 1940
- [Background] Houston WJ. The analysis of errors in orthodontic measurements. Am J Orthod. 1983 May;83(5):382-90. doi: 10.1016/0002-9416(83)90322-6. PMID 6573846
- [Background] Moynihan PJ. The role of diet and nutrition in the etiology and prevention of oral diseases. Bull World Health Organ. 2005 Sep;83(9):694-9. Epub 2005 Sep 30. PMID 16211161
- [Background] Manfred L, Covell DA, Crowe JJ, Tufekci E, Mitchell JC. A novel biomimetic orthodontic bonding agent helps prevent white spot lesions adjacent to brackets. Angle Orthod. 2013 Jan;83(1):97-103. doi: 10.2319/110811-689.1. Epub 2012 Jun 27. PMID 22765388
- [Background] Gizani S, Petsi G, Twetman S, Caroni C, Makou M, Papagianoulis L. Effect of the probiotic bacterium Lactobacillus reuteri on white spot lesion development in orthodontic patients. Eur J Orthod. 2016 Feb;38(1):85-89. doi: 10.1093/ejo/cjv015. Epub 2015 Apr 3. PMID 25840585
- [Background] Julien KC, Buschang PH, Campbell PM. Prevalence of white spot lesion formation during orthodontic treatment. Angle Orthod. 2013 Jul;83(4):641-7. doi: 10.2319/071712-584.1. Epub 2013 Jan 4. PMID 23289733
- [Background] van Loveren C, Duggal MS. The role of diet in caries prevention. Int Dent J. 2001;51(6 Suppl 1):399-406. doi: 10.1111/j.1875-595x.2001.tb00586.x. PMID 11794561
- [Background] Stookey GK. The effect of saliva on dental caries. J Am Dent Assoc. 2008 May;139 Suppl:11S-17S. doi: 10.14219/jada.archive.2008.0347. PMID 18595200
- [Background] Keller MK, Nohr Larsen I, Karlsson I, Twetman S. Effect of tablets containing probiotic bacteria (Lactobacillus reuteri) on early caries lesions in adolescents: a pilot study. Benef Microbes. 2014 Dec;5(4):403-7. doi: 10.3920/BM2013.0089. PMID 24889893
- [Background] Talaat, D. Effect of Probiotic Chewable Tablets on Oral Health and White Spot Lesions in Pre-school Children: A Randomized Clinical Trial. Egypt Dent J. 2021; 67: 1797-1807.
- [Background] Flichy-Fernandez AJ, Ata-Ali J, Alegre-Domingo T, Candel-Marti E, Ata-Ali F, Palacio JR, Penarrocha-Diago M. The effect of orally administered probiotic Lactobacillus reuteri-containing tablets in peri-implant mucositis: a double-blind randomized controlled trial. J Periodontal Res. 2015 Dec;50(6):775-85. doi: 10.1111/jre.12264. Epub 2015 Feb 25. PMID 25712760